CLINICAL TRIAL: NCT06943430
Title: The Effect of Laughter Yoga Applied to Nursing Students on Exam Anxiety and Spirituality
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Hande Tiftikci, Student Principal Investigator(Under Supervision of Prof. Dr. Hüsna Özveren, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KKU-SBF-HT-01
Record Dates: First submitted 2025-04-10; First posted 2025-04-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Exam Stress; Anxiety; Spirituality
Keywords: laughter yoga; exam stress; anxiety; spirituality
MeSH Terms: conditions — Anxiety Disorders | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, the data were entered by someone other than the researcher, and statistical analysis was performed by a person other than the researcher. In the study, laughter yoga was applied to the participants in the experimental group. Since laughter yoga is an intervention that can be clearly recognized by the participants, they were aware of which group they were in. This means that blinding of the participants was not possible. Additionally, since the researcher was the person implementing the intervention, both the participants and the researcher were aware of the intervention. Therefore, blinding was not included in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Participants in the intervention group received laughter yoga sessions twice a week for a total of four weeks.
  Interventions: Other: laughter yoga
- Control (No Intervention): No application was made to the control group, standard procedure was followed.

INTERVENTIONS:
Other: laughter yoga — Participants in the intervention group received laughter yoga sessions twice a week for a total of four weeks.
  Arms: intervention

SUMMARY:
This study is planned as a randomized controlled trial to determine the effect of laughter yoga on the exam anxiety and spirituality levels of nursing students. The research will be conducted with 100 second-year nursing students between 04.2025 and 06.2025. Students who meet the inclusion criteria will be randomized and divided into two groups: the experimental group (n=36) and the control group (n=36). All participating students will be administered the "Demographic Characteristics Form," "Exam Anxiety Scale," and "Spirituality Scale" (pre-test).

The experimental group will undergo laughter yoga sessions twice a week for 4 weeks, totaling 8 sessions.

The control group will only complete the "Demographic Characteristics Form," "Exam Anxiety Scale," and "Spirituality Scale" (pre-test). No intervention will be applied to the control group.

After the laughter yoga sessions are completed, both the experimental and control groups will complete the "Demographic Characteristics Form," "Exam Anxiety Scale," and "Spirituality Scale" (post-test).

The collected data will be analyzed using SPSS 22 software.

DETAILED DESCRIPTION:
Research Hypotheses:

Laughter yoga reduces exam anxiety in nursing students. Laughter yoga increases the spirituality levels of nursing students. This research aims to examine the effects of laughter yoga on exam anxiety and spirituality levels in nursing students. The researcher has completed a two-day "Laughter Yoga Leader" training with an Internationally Certified Laughter Yoga Instructor and has received the "Laughter Yoga Trainer Training" certificate. The study was conducted with an experimental design, including an experimental group and a control group. The interventions were applied by the researcher, who holds the "Laughter Yoga Leader" certification.

The sample was selected using the simple random sampling method, and participants were initially administered the "Demographic Information Form," "Exam Anxiety Scale," and "Spirituality Scale." After obtaining ethical committee approval, laughter yoga sessions were applied to students in the experimental group, while no intervention was provided to the control group. As the study was designed experimentally, both groups were initially evaluated using the same measurement tools, and then the experimental group underwent laughter yoga sessions. After the laughter yoga sessions, data were collected from both groups using the same measurement tools, and changes in exam anxiety and spirituality levels were analyzed.

The collected data were evaluated to analyze the changes in exam anxiety and spirituality levels. This study aims to determine the effects of laughter yoga on reducing exam anxiety and increasing spirituality levels in nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Being a 2nd-year student in the Nursing Department
* Able to speak and understand Turkish
* Voluntarily agreeing to participate in the study
* No visual or hearing impairments
* No history of psychiatric illness
* No current or past use of psychotropic medication

Exclusion Criteria:

* Refusal to participate in the study
* Inability to speak or understand Turkish
* Diagnosed psychiatric illness and/or use of psychotropic agents
* Previous participation in laughter yoga
* Physical limitations or respiratory problems preventing yoga practice
* Difficulty in performing breathing exercises due to conditions such as septum deviation
* Abdominal surgery within the past 6 months

Drop-out Criteria:

* Failure to attend any of the laughter yoga sessions
* Receiving a new diagnosis that contraindicates laughter yoga during the 4-week intervention period

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-04-27 (Estimated); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
Change in exam anxiety levels as measured by the Test Anxiety Scale | Baseline and post-intervention (Week 4)
  Exam anxiety will be assessed using a validated Test Anxiety Scale before and after the 4-week laughter yoga intervention.
  The mean score difference between pre-test and post-test will be analyzed using paired samples t-test.

SECONDARY OUTCOMES:
Change in spirituality levels as measured by the Spirituality Scale | Baseline and post-intervention (Week 4)
  Spirituality levels will be measured using a validated Spirituality Scale at the beginning and end of the intervention.
  Differences in mean scores will be analyzed with paired t-tests to determine statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Tiftikci, Principal Investigator — Kırıkkale University
Locations (1):
- Kirikkale University, Kırıkkale, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The confidentiality of the data used in the study will be protecte